CLINICAL TRIAL: NCT03834545
Title: Improvement of Motivation for Physical Activity in an Institutionalized Geriatric Population Thanks to a Virtual Environment: Comparison of Motivation Between Classic Bike and Bike With Virtual Environment
Brief Title: Improved Motivation for Physical Activity in an Institutionalized Geriatric Population Through a Virtual Environment
Acronym: Cyclepad Pilot
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: ARUET
Record Dates: First submitted 2019-01-30; First posted 2019-02-08 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2019-02

CONDITIONS: Motivation; Fall

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cycling group: They attended three sessions of exercise on three different conditions : a classic ergometric bicycle without chairback, an ergometric bicycle with chairback with virtual environment and the other session without virtual environment

SUMMARY:
The purpose of this study is to test the interest of a virtual environment with cycling to increase the motivation of physical activity practice in institutionalized older adults.

DETAILED DESCRIPTION:
The World Health Organization (WHO) recommends for people aged 65 years and over a weekly practice of at least 150 minutes of moderate-intensity endurance activities or at least 75 minutes of activity. endurance of sustained intensity, or an equivalent combination of moderate and sustained activity. However, the attractiveness for physical activity fades over the years limiting the practice of physical activity. Several types of unconventional approaches have already shown their effectiveness in the prevention of falls in the elderly but these practices find their limits in the lack of adherence to this type of exercise, especially in nursing homes. New virtual reality and gaming technologies have recently emerged and are being used as tools to prevent the risk of falling. The use of these new tools has advantages over conventional exercises: motivating.

The investigators aimed to test the interest of a virtual environment with cycling to increase the motivation of physical activity practice in institutionalized older adults.

ELIGIBILITY:
Inclusion Criteria:

* age over 65
* ability to cycle

Exclusion Criteria:

* unstable cardiopathy
* New York Heart Association classification III or IV
* severe cognitive disorders with inability to follow simple orders (follow investigator, ride on the ergometric bicycles, pedal)
* visual disturbance preventing counting fingers at 5m

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Institutionalized older adults over 65 years
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Cycling distance in meters | 3 months
  Primary outcome was the cycling distance measured at each session without encouragement

SECONDARY OUTCOMES:
Time spent pedaling in seconds per session | 3 months
  Measure of the time spent pedaling per session without encouragement
The average speed in meters per second per session | 3 months
  Measure of the average cycling speed per session without encouragement.
Mean pedaling cadence per session in revolutions per minute | 3 months
  Measure of the average pedaling cadence per session without encouragement.
Borg rating of perceived exertion scale | 3 months
  Measure of the perceived exertion after each cycling session with Borg rating of perceived exertion scale. Range 0-10. Ten corresponding to the maximal perceived exertion
Mean pedaling power per session in Watts | 3 months
  Measure of the pedaling power per session without encouragement
Closed-ended question to know which condition they would prefer for a futur exercise session. | 3 months
  Participant were asked at the end of the third session, which condition they would prefer for a futur exercice session. Possible answers: "Classic ergometric bicycle Kettler E3)", "Cycleo without virtual environment", "Cycleo with virtual environment", "None".

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Normandy, France

IPD SHARING:
Plan to Share IPD: Undecided